CLINICAL TRIAL: NCT05766527
Title: A Phase 1 Safety and Tolerability Study of KM602 in Patients With Advanced Solid Tumors
Brief Title: A Study of KM602 in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM602-1001
Record Dates: First submitted 2023-02-28; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KM602 monotherapy (Experimental): Dose escalation and expansion
  Interventions: Biological: KM602

INTERVENTIONS:
Biological: KM602 — Multiple dose levels of KM602 will be administered, including 0.01 mg/kg QW, 0.1 mg/kg QW, 0.6 mg/kg QW, 3 mg/kg QW, and 10 mg/kg QW. KM602 is administered intravenously once a week, and each cycle is 21 days.

SUMMARY:
This study is a Phase 1 open-label, first-in-human, multicenter study to evaluate the safety, tolerability, pharmacokinetics, and activity of KM602 as monotherapy in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This Phase 1 study is comprised of dose escalation and expansions for KM602 monotherapy. Monotherapy dose escalation is designed with initial accelerated titration followed by a standard 3+3 dose escalation; Patients will remain on study treatment until progression of disease, unacceptable toxicity, or other specified reason for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, disease that is unresectable, locally advanced, or metastatic and has progressed following all standard treatments or is not appropriate for standard treatments (predominantly melanoma and non-small cell lung cancer)
2. All patients must have at least one measurable lesion at baseline according to RECIST v1.1
3. ECOG performance status of 0 or 1
4. Life expectancy of ≥ 12 weeks
5. Adequate baseline hematologic, renal, and hepatic function

Exclusion Criteria:

1. Patients with meningeal metastasis or symptomatic central nervous system metastasis
2. Any second malignancy active within the previous 5 years
3. Any active, known, or suspected autoimmune disease
4. Active or prior pneumonitis or interstitial lung disease
5. Prior organ allograft or allogeneic hematopoietic stem cell transplantation
6. Treatment with any anti-cancer therapy or participation in another investigational drug or biologics trial within 4 weeks prior to the first dose of KM602
7. Prior treatment with a CTLA-4 antagonist, including ipilimumab and tremelimumab
8. History of ≥ Grade 3 immune-related adverse event leading to treatment discontinuation
9. Systemic treatment with corticosteroids (> 10 mg/day prednisone) or other immunosuppressive medication within 14 days prior to the first dose of KM602 or during the study
10. Known seropositivity for or active infection by human immunodeficiency virus, hepatitis B or C
11. Known allergies, hypersensitivity, or intolerance to KM602 or excipients in the drug product formulation
12. Active infection requiring therapy at the time of the first dose of KM602
13. Pregnancy or breastfeeding
14. Any serious or uncontrolled health condition, which, in the opinion of the Investigator, would place the subject at undue risk from the study, impair the ability of the subject to receive protocol specified therapy, or interfere with the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of KM602, if any | Approximately 15 months
  Determined by the frequency of dose-limiting toxicities during dose-escalation
Recommended Phase 2 dose (RP2D) of KM602 | Approximately 15 months
  Determined by the frequency of dose-limiting toxicities during dose-escalation
Incidence of treatment emergent adverse events | Through study completion, approximately 28 months
  Severity graded per CTCAE version 5.0

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of KM602 | Through study completion, approximately 28 months
Area Under the Curve (AUC) of KM602 | Through study completion, approximately 28 months
t1/2 of KM602 | Through study completion, approximately 28 months
Plasma clearance (CL) of KM602 | Through study completion, approximately 28 months
Volume of distribution (V) of KM602 | Through study completion, approximately 28 months
Anti-Drug Antibody of KM602 | Through study completion, approximately 28 months
Objective Response Rate (ORR) of KM602 | Through study completion, approximately 28 months
Disease Control Rate (DCR) of KM602 | Through study completion, approximately 28 months
Progression-free survival(PFS) of KM602 | Through study completion, approximately 28 months
Duration of Response (DOR) of KM602 | Through study completion, approximately 28 months
Overall survival (OS) of KM602 | Through study completion, approximately 28 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China